CLINICAL TRIAL: NCT04529395
Title: Impact of Aromatherapy on the Delirium of Patients in Intensive Care Unit
Acronym: AROMADELI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GHRMSA 1017; IDRCB 2019-A01978-49 (Other: ANSM)
Record Dates: First submitted 2020-08-03; First posted 2020-08-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2023-10

CONDITIONS: Intensive Care Unit Delirium
Keywords: Intensive Care Unit; Delirium; Aromatherapy
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy group (Experimental)
  Interventions: Other: Blending of essential oils
- Control group (Active Comparator)
  Interventions: Other: Apricot vegetable oil

INTERVENTIONS:
Other: Blending of essential oils — The mixture of essential oils will be applied to the arch of the foot by massage every 8 hours (3 times a day, 6 drops per application with 3 drops per foot).
  Arms: Aromatherapy group
Other: Apricot vegetable oil — The apricot vegetable oil will be applied to the arch of the foot by massage every 8 hours (3 times a day, 6 drops per application with 3 drops per foot).
  Arms: Control group

SUMMARY:
The primary objective of this monocenter randomized controlled trial is to assess the efficacy of aromatherapy to prevent delirium in patients hospitalized in an intensive care unit.

DETAILED DESCRIPTION:
Secondary objectives:

1. To assess the efficacy of aromatherapy on :

   * the level of consciousness,
   * pain,
   * the duration of mechanical ventilation,
   * the occurence of an accidental extubation,
   * the length of stay in the intensive care unit,
   * the cumulative duration of delirium episodes,
   * the time until first episode of delirium,
   * the use of neuroleptics.
2. To determine the factors influencing the efficacy of aromatherapy.
3. To assess the safety of aromatherapy.

Conduct of research:

After inclusion, patients will be randomized between the aromatherapy and control groups. Treatment will be started on the same day as randomization.

Aromatherapy treatment will consist of a dermal application on the feet of a mixture of essential oils.

Control treatment will consist of a dermal application on the feet of apricot vegetable oil.

The mixture of essential oils (aromatherapy group) or vegetable oil (control group) will be applied to the arch of the foot by massage, every eight hours, at a rate of six drops per application (3 drops per foot).

Treatment will continue until the patient is discharged from the intensive care unit or no later than 15 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient hospitalized in an intensive care unit for an expected duration of at least 24 hours
* Patient requiring mechanical ventilation with initial therapeutic sedation adapted secondarily for comfort sedation, defined by a RASS score target between -2 and 0
* Patient affiliated to/beneficiary of a social security scheme

Exclusion Criteria:

* Allergy to essential and/or vegetable oils
* Palliative sedation
* Foot skin injury contraindicating the application of an oil
* Moribund patient or expected death
* History of dementia
* Participation to a RIPH-1 study
* Pregnant or breastfeeding woman
* Patient under legal protection
* Patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of delirium | Up to 15 days after randomization
  The occurrence of delirium will be defined by the presence of at least one episode during the patient's stay in the intensive care unit, diagnosed using the CAM-ICU scale.

SECONDARY OUTCOMES:
Score on the Richmond Agitation-Sedation Scale | Up to 15 days after randomization
Score on the Behavior-Pain Scale | Up to 15 days after randomization
Duration of mechanical ventilation between admission and first extubation | Up to 15 days after randomization
Occurrence of at least one accidental extubation during the stay | Up to 15 days after randomization
Length of stay in intensive care unit | Up to 15 days after randomization
Cumulative duration of delirium episodes | Up to 15 days after randomization
Time until first episode of delirium | Up to 15 days after randomization
Duration of neuroleptic treatment | Up to 15 days after randomization
Occurrence of a local allergic reaction | Up to 15 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Kuteifan, MD, Principal Investigator — GHRMSA hospital
Locations (1):
- Groupe Hospitalier de Mulhouse et de la Région Sud-Alsace, Mulhouse, France

IPD SHARING:
Plan to Share IPD: No